CLINICAL TRIAL: NCT00942292
Title: Randomised Controlled Trial of the Effects of Fish Oil Emulsion in Total Parenteral Nutrition Upon Tumour Vascularity in Patients With Hepatic Colorectal Metastases
Brief Title: The Effect of Fish Oils on Human Hepatic Colorectal Metastases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Collaborators: B. Braun Melsungen AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: 10097; REC reference: 06/Q2501/160; EudraCT number: 2006-000044-71
Record Dates: First submitted 2009-07-16; First posted 2009-07-20 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Colorectal Liver Metastases
Keywords: Hepatic; colorectal; metastases; TPN; Fish oil
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lipidem (fish oil) (Active Comparator): Lipidem (TPN containing fish oil)
  Interventions: Dietary Supplement: Lipidem- fish oil emulsion BBraun UK; Procedure: Digital Contrast MRI scan
- Lipofundin (TPN) (Active Comparator): Control arm (no fish oil)
  Interventions: Dietary Supplement: Lipidem- fish oil emulsion BBraun UK; Procedure: Digital Contrast MRI scan

INTERVENTIONS:
Dietary Supplement: Lipidem- fish oil emulsion BBraun UK
Procedure: Digital Contrast MRI scan

SUMMARY:
The purpose of this study is to determine whether fish oils - a known source of omega-3 given intravenously (via a 'drip') will help cure secondary deposits in the liver from bowel cancer.

DETAILED DESCRIPTION:
Fish oils have many proven benefits for a wide range of clinical arenas such as ischaemic heart disease, rheumatoid arthritis and inflammatory bowel disease.

Recent research has described the beneficial effects of intravenous fish oils for surgical patients, such as reduced hospital stay, reduced re-operation rate and reduced requirements for intravenous antibiotics. These are in part due to the anti-inflammatory effects of fish oils.

There is evidence that fish oils are also effective against cancer, large population studies indicate that diets rich in omega-3 are associated with a lower incidence of cancer, and in vitro and animal studies demonstrate anti-tumour effects of fish oils

1. Fish oils inhibit the growth of different human cancer cell lines
2. They act specifically on tumour cells only and do not impair the function of normal cells
3. EPA and DHA inhibit the growth of human cancer cell lines and enhance apoptosis.
4. Fish oil induces apoptosis in human colorectal cancer cell lines in-vitro after 48hrs incubation
5. Fish oil has been shown to inhibit the proliferation activities, inhibit the invasive activities and increase the apoptosis of human pancreatic carcinoma cell lines in-vitro after only 48hrs of exposure
6. Fish oil has been shown to enhance colorectal adenocarcinoma cell lines sensitivity to radiotherapy
7. Fish oil has also been shown to reduce the incidence of liver metastases in experimentally induced ductal pancreatic cancer in rats after 30 weeks of oral treatment with an omega-3 supplemented diet.
8. Lung cancer xenografts in animals fed with fish oil showed significantly increased tumour regression in response to doxorubicin compared to those fed with omega-3.

This study aims to assess the effect of omega-3 FA upon hepatic colorectal metastases in a pilot study. 20 patients will be selected for this pilot study with potentially resectable hepatic colorectal adenocarcinoma metastases. 10 patients will receive total parenteral nutrition (TPN) without fish oils (controls), 10 will receive fish oil containing lipid emulsion in their TPN.

Changes in tumour angiogenesis (increased angiogenesis is associated with a poorer prognosis in hepatic colorectal metastases) will be investigated using digital contrast enhanced MRI scanning, and markers of angiogenesis will be investigated in blood and resected tumour samples from the patients.

It is a randomised controlled double blind trial.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-80
2. Able to give informed written consent
3. Diagnosis of respectable hepatic colorectal metastases on radiological and laparoscopic appearances

Exclusion Criteria:

1. Patients already taking fish oil supplements
2. Hypersensitivity to fish-, egg-, or soy protein, or to any of the active substances or constituents in the lipid emulsion
3. Hyperlipidaemia
4. Severe blood coagulation disorders
5. Severe renal insufficiency (Creatinine >200)
6. Any general contra-indications to infusion therapy - pulmonary oedema, hyperhydration, decompensated cardiac insufficiency
7. Any unstable medical conditions - uncontrolled diabetes mellitus, acute myocardial infarction, stroke, embolic disease, metabolic acidosis, sepsis, pancreatitis
8. Patients undergoing conventional neo-adjuvant chemotherapy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2007-05; Primary Completion 2009-12 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Change in gadolinium chelate enhancement on DCE-MRI between study entry and exit, as determined by calculating the bi-directional transfer co-efficient.(Changes in tumour angiogenesis after treatment with fish oils or control TPN) | 72 hours

SECONDARY OUTCOMES:
Changes in biomarkers of inflammation and angiogenesis in the patient's blood and resected tumour samples | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Ashley R Dennison, MBChB, FRCS, MD, Principal Investigator — Leicester General Hospital
Locations (1):
- Leicester General Hospital, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Background] Morlion BJ, Torwesten E, Lessire H, Sturm G, Peskar BM, Furst P, Puchstein C. The effect of parenteral fish oil on leukocyte membrane fatty acid composition and leukotriene-synthesizing capacity in patients with postoperative trauma. Metabolism. 1996 Oct;45(10):1208-13. doi: 10.1016/s0026-0495(96)90237-1. PMID 8843174
- [Background] Roulet M, Frascarolo P, Pilet M, Chapuis G. Effects of intravenously infused fish oil on platelet fatty acid phospholipid composition and on platelet function in postoperative trauma. JPEN J Parenter Enteral Nutr. 1997 Sep-Oct;21(5):296-301. doi: 10.1177/0148607197021005296. PMID 9323693
- [Background] Schauder P, Rohn U, Schafer G, Korff G, Schenk HD. Impact of fish oil enriched total parenteral nutrition on DNA synthesis, cytokine release and receptor expression by lymphocytes in the postoperative period. Br J Nutr. 2002 Jan;87 Suppl 1:S103-10. doi: 10.1079/bjn2001463. PMID 11895146
- [Background] Mayer K, Fegbeutel C, Hattar K, Sibelius U, Kramer HJ, Heuer KU, Temmesfeld-Wollbruck B, Gokorsch S, Grimminger F, Seeger W. Omega-3 vs. omega-6 lipid emulsions exert differential influence on neutrophils in septic shock patients: impact on plasma fatty acids and lipid mediator generation. Intensive Care Med. 2003 Sep;29(9):1472-81. doi: 10.1007/s00134-003-1900-2. Epub 2003 Jul 25. PMID 12897994
- [Background] Mayer K, Gokorsch S, Fegbeutel C, Hattar K, Rosseau S, Walmrath D, Seeger W, Grimminger F. Parenteral nutrition with fish oil modulates cytokine response in patients with sepsis. Am J Respir Crit Care Med. 2003 May 15;167(10):1321-8. doi: 10.1164/rccm.200207-674OC. Epub 2003 Feb 25. PMID 12615625
- [Background] Schulzki, C., et al., Effect of a new type of lipid emulsion base on soybean oil, MCT, olive oil and fish oil (SMOF) in surgical patients. Clinical Nutrition, 1999. 19(Supp 1): p. S7.
- [Background] Weiss G, Meyer F, Matthies B, Pross M, Koenig W, Lippert H. Immunomodulation by perioperative administration of n-3 fatty acids. Br J Nutr. 2002 Jan;87 Suppl 1:S89-94. doi: 10.1079/bjn2001461. PMID 11895158
- [Background] Grimminger, F., W. Seeger, and K. Mayer, Use of omeg-3 fatty acid-containing lipid emulsions in the intensive care unit environment: the clinician's view. Clinical Nutrition, 2002. 21(2): p. 23-9.
- [Background] Grimble, R., et al., Effects of fish oil supplementation on ability of monocytes to invoke a pro-inflammatory response in endothelial cells. Clinical Nutrition, 2004. 23(4): p. 833-834.
- [Background] Morlion, B., et al., What is the optimum omega-3 to omega-6 fatty acid (FA) ratio of patenteral lipid emulsions in post-operative trauma? Clinical Nutrition, 1997. 16(Suppl 2): p. 49.
- [Background] Furst P, Kuhn KS. Fish oil emulsions: what benefits can they bring? Clin Nutr. 2000 Feb;19(1):7-14. doi: 10.1054/clnu.1999.0072. No abstract available. PMID 10700528
- [Background] Adolph, M., Lipid emulsions in parenteral nutrition - state of the art and future perspectives. Clinical Nutrition, 2001. 20(Suppl 4): p. 1
- [Background] Grimm H, Tibell A, Norrlind B, Blecher C, Wilker S, Schwemmle K. Immunoregulation by parenteral lipids: impact of the n-3 to n-6 fatty acid ratio. JPEN J Parenter Enteral Nutr. 1994 Sep-Oct;18(5):417-21. doi: 10.1177/0148607194018005417. PMID 7815672
- [Background] Grimm H, Kraus A. Immunonutrition--supplementary amino acids and fatty acids ameliorate immune deficiency in critically ill patients. Langenbecks Arch Surg. 2001 Aug;386(5):369-76. doi: 10.1007/s004230100241. PMID 11685569
- [Background] Grecu, I., L. Mirea, and I. Grintescu, Parenteral fish oil supplementation in patients with abdominal sepsis. Clinical Nutrition, 2003. 22: p. S23
- [Background] Heller, A., J. Striebel, and T. Koch, Effects of fish-oil supplementation on the clinical course of critical illness. A multicenter trial. European Journal of Anesthesiology, 2003. 20: p. 157.
- [Background] Tsekos E, Reuter C, Stehle P, Boeden G. Perioperative administration of parenteral fish oil supplements in a routine clinical setting improves patient outcome after major abdominal surgery. Clin Nutr. 2004 Jun;23(3):325-30. doi: 10.1016/j.clnu.2003.07.008. PMID 15158295
- [Background] Kelbel, I., et al., Effects of omega-3 fatty acids on immune function: a double-blind, randomized trial of fish oil based infusion in post-operative patients. Clinical Nutrition, 2002. 21: p. 13-14.
- [Background] Wichmann, M., et al., Reduction of length of post-operative stay by fish oil containing lipid emulsion - data from a multicenter trial. Clinical Nutrition, 2004. 23
- [Background] Heller AR, Rossel T, Gottschlich B, Tiebel O, Menschikowski M, Litz RJ, Zimmermann T, Koch T. Omega-3 fatty acids improve liver and pancreas function in postoperative cancer patients. Int J Cancer. 2004 Sep 10;111(4):611-6. doi: 10.1002/ijc.20291. PMID 15239141
- [Background] Llor, X., et al., Involvement of the intrinsic and extrinsic pathways in the apoptosis-inducing effect of the n-3 fatty acid docosahexanoic on colorectal cancer cells. Clinical Nutrition, 2004. 23(4): p. 891.
- [Background] Shirota, T., et al., Suppression of human pancreatic carcinoma cell growth and invasion by eicosapentaenoic acid. Clinical Nutrition, 2004. 23(4): p. 888-889
- [Background] Jiang YH, Lupton JR, Chang WC, Jolly CA, Aukema HM, Chapkin RS. Dietary fat and fiber differentially alter intracellular second messengers during tumor development in rat colon. Carcinogenesis. 1996 Jun;17(6):1227-33. doi: 10.1093/carcin/17.6.1227. PMID 8681436
- [Background] Singh J, Hamid R, Reddy BS. Dietary fat and colon cancer: modulation of cyclooxygenase-2 by types and amount of dietary fat during the postinitiation stage of colon carcinogenesis. Cancer Res. 1997 Aug 15;57(16):3465-70. PMID 9270014
- [Background] Chen ZY, Istfan NW. Docosahexaenoic acid is a potent inducer of apoptosis in HT-29 colon cancer cells. Prostaglandins Leukot Essent Fatty Acids. 2000 Nov;63(5):301-8. doi: 10.1054/plef.2000.0218. PMID 11090257
- [Background] Narayanan BA, Narayanan NK, Reddy BS. Docosahexaenoic acid regulated genes and transcription factors inducing apoptosis in human colon cancer cells. Int J Oncol. 2001 Dec;19(6):1255-62. doi: 10.3892/ijo.19.6.1255. PMID 11713597
- [Background] Chiu LC, Wan JM. Induction of apoptosis in HL-60 cells by eicosapentaenoic acid (EPA) is associated with downregulation of bcl-2 expression. Cancer Lett. 1999 Oct 18;145(1-2):17-27. doi: 10.1016/s0304-3835(99)00224-4. PMID 10530765
- [Background] Collett ED, Davidson LA, Fan YY, Lupton JR, Chapkin RS. n-6 and n-3 polyunsaturated fatty acids differentially modulate oncogenic Ras activation in colonocytes. Am J Physiol Cell Physiol. 2001 May;280(5):C1066-75. doi: 10.1152/ajpcell.2001.280.5.C1066. PMID 11287318
- [Background] Dommels YE, Alink GM, Linssen JP, van Ommen B. Effects of n-6 and n-3 polyunsaturated fatty acids on gap junctional intercellular communication during spontaneous differentiation of the human colon adenocarcinoma cell line Caco-2. Nutr Cancer. 2002;42(1):125-30. doi: 10.1207/S15327914NC421_17. PMID 12235644
- [Background] Wenger, F., et al., Impact of dietary fact on hepatic metastases and lipidperoxidation in pancreatic cancer. Clinical Nutrition, 2004. 23(4): p. 788-789.
- [Background] Saeki T, Tanada M, Takashima S, Saeki H, Takiyama W, Nishimoto N, Moriwaki S. Correlation between expression of platelet-derived endothelial cell growth factor (thymidine phosphorylase) and microvessel density in early-stage human colon carcinomas. Jpn J Clin Oncol. 1997 Aug;27(4):227-30. doi: 10.1093/jjco/27.4.227. PMID 9379508
- [Background] O'Reilly MS, Boehm T, Shing Y, Fukai N, Vasios G, Lane WS, Flynn E, Birkhead JR, Olsen BR, Folkman J. Endostatin: an endogenous inhibitor of angiogenesis and tumor growth. Cell. 1997 Jan 24;88(2):277-85. doi: 10.1016/s0092-8674(00)81848-6. PMID 9008168
- [Background] Rose DP, Connolly JM. Omega-3 fatty acids as cancer chemopreventive agents. Pharmacol Ther. 1999 Sep;83(3):217-44. doi: 10.1016/s0163-7258(99)00026-1. PMID 10576293
- [Background] Benais-Pont, G., Y. Dupertuis, and C. Pichard, Influence of polyunsaturated fatty acids on the growth and radio-sensitivity of three human colorectal adenocarcinoma cell lines. Clinical Nutrition, 2004. 23(4): p. 801
- [Background] Sturlan, S., et al., Long-chain omega-3 polyunsaturated fatty acids enhance arsenic trioxide cytotoxicity in breast cancer cells. Clinical Nutrition, 2004. 23(4): p. 797
- [Background] Heller AR, Fischer S, Rossel T, Geiger S, Siegert G, Ragaller M, Zimmermann T, Koch T. Impact of n-3 fatty acid supplemented parenteral nutrition on haemostasis patterns after major abdominal surgery. Br J Nutr. 2002 Jan;87 Suppl 1:S95-101. doi: 10.1079/bjn2001462. PMID 11895160
- [Background] Katz DP, Manner T, Furst P, Askanazi J. The use of an intravenous fish oil emulsion enriched with omega-3 fatty acids in patients with cystic fibrosis. Nutrition. 1996 May;12(5):334-9. doi: 10.1016/s0899-9007(96)80056-6. PMID 8875517
- [Background] Tappy, L., et al., Metabolic effects of parenteral nutrition with or without omega-3 fatty acids. Clinical Nutrition, 2003. 22: p. S50.
- [Background] Mertes N, Grimm H, Furst P, Stehle P. Safety and efficacy of a new parenteral lipid emulsion (SMOFlipid) in surgical patients: a randomized, double-blind, multicenter study. Ann Nutr Metab. 2006;50(3):253-9. doi: 10.1159/000091683. Epub 2006 Feb 23. PMID 16508253
- [Background] Genton, L., et al., Tolerance to a lipid emulsion containing a mixture of soybean, olive, coconut and fish oils compared with a standard fat emulsion containing only soybean oil. Clinical Nutrition, 2004. Abstract ESPEN 2004.
- [Background] Antebi H, Mansoor O, Ferrier C, Tetegan M, Morvan C, Rangaraj J, Alcindor LG. Liver function and plasma antioxidant status in intensive care unit patients requiring total parenteral nutrition: comparison of 2 fat emulsions. JPEN J Parenter Enteral Nutr. 2004 May-Jun;28(3):142-8. doi: 10.1177/0148607104028003142. PMID 15141405
- [Background] Mayer K, Meyer S, Reinholz-Muhly M, Maus U, Merfels M, Lohmeyer J, Grimminger F, Seeger W. Short-time infusion of fish oil-based lipid emulsions, approved for parenteral nutrition, reduces monocyte proinflammatory cytokine generation and adhesive interaction with endothelium in humans. J Immunol. 2003 Nov 1;171(9):4837-43. doi: 10.4049/jimmunol.171.9.4837. PMID 14568963
- [Background] Schlotzer, E., et al., Intravenous application of a fish oil emulsion. Akt Ernahr Med, 1992. 17: p. 170-5.
- [Background] Richelle, M., et al., Does fish oil supplementation effect the intravascular effect of LCT emulsion in man. Clinical Nutrition, 1993: p. 12.
- [Background] Moertel CG, Hanley JA. The effect of measuring error on the results of therapeutic trials in advanced cancer. Cancer. 1976 Jul;38(1):388-94. doi: 10.1002/1097-0142(197607)38:13.0.co;2-a. PMID 947531
- [Background] James K, Eisenhauer E, Christian M, Terenziani M, Vena D, Muldal A, Therasse P. Measuring response in solid tumors: unidimensional versus bidimensional measurement. J Natl Cancer Inst. 1999 Mar 17;91(6):523-8. doi: 10.1093/jnci/91.6.523. PMID 10088622
- [Background] Yuh WT. An exciting and challenging role for the advanced contrast MR imaging. J Magn Reson Imaging. 1999 Sep;10(3):221-2. doi: 10.1002/(sici)1522-2586(199909)10:33.0.co;2-x. No abstract available. PMID 10508280
- [Background] Taylor JS, Tofts PS, Port R, Evelhoch JL, Knopp M, Reddick WE, Runge VM, Mayr N. MR imaging of tumor microcirculation: promise for the new millennium. J Magn Reson Imaging. 1999 Dec;10(6):903-7. doi: 10.1002/(sici)1522-2586(199912)10:63.0.co;2-a. PMID 10581502
- [Background] Buadu LD, Murakami J, Murayama S, Hashiguchi N, Sakai S, Masuda K, Toyoshima S, Kuroki S, Ohno S. Breast lesions: correlation of contrast medium enhancement patterns on MR images with histopathologic findings and tumor angiogenesis. Radiology. 1996 Sep;200(3):639-49. doi: 10.1148/radiology.200.3.8756909.
- [Background] Hawighorst H, Knapstein PG, Weikel W, Knopp MV, Zuna I, Knof A, Brix G, Schaeffer U, Wilkens C, Schoenberg SO, Essig M, Vaupel P, van Kaick G. Angiogenesis of uterine cervical carcinoma: characterization by pharmacokinetic magnetic resonance parameters and histological microvessel density with correlation to lymphatic involvement. Cancer Res. 1997 Nov 1;57(21):4777-86. PMID 9354439
- [Background] Hawighorst H, Weikel W, Knapstein PG, Knopp MV, Zuna I, Schonberg SO, Vaupel P, van Kaick G. Angiogenic activity of cervical carcinoma: assessment by functional magnetic resonance imaging-based parameters and a histomorphological approach in correlation with disease outcome. Clin Cancer Res. 1998 Oct;4(10):2305-12. PMID 9796959
- [Background] Mayr NA, Hawighorst H, Yuh WT, Essig M, Magnotta VA, Knopp MV. MR microcirculation assessment in cervical cancer: correlations with histomorphological tumor markers and clinical outcome. J Magn Reson Imaging. 1999 Sep;10(3):267-76. doi: 10.1002/(sici)1522-2586(199909)10:33.0.co;2-y. PMID 10508286
- [Background] Erlemann R, Sciuk J, Bosse A, Ritter J, Kusnierz-Glaz CR, Peters PE, Wuisman P. Response of osteosarcoma and Ewing sarcoma to preoperative chemotherapy: assessment with dynamic and static MR imaging and skeletal scintigraphy. Radiology. 1990 Jun;175(3):791-6. doi: 10.1148/radiology.175.3.2188300.
- [Background] Fletcher BD, Hanna SL, Fairclough DL, Gronemeyer SA. Pediatric musculoskeletal tumors: use of dynamic, contrast-enhanced MR imaging to monitor response to chemotherapy. Radiology. 1992 Jul;184(1):243-8. doi: 10.1148/radiology.184.1.1319075.
- [Background] Reddick WE, Taylor JS, Fletcher BD. Dynamic MR imaging (DEMRI) of microcirculation in bone sarcoma. J Magn Reson Imaging. 1999 Sep;10(3):277-85. doi: 10.1002/(sici)1522-2586(199909)10:33.0.co;2-s. PMID 10508287
- [Background] Barentsz JO, Berger-Hartog O, Witjes JA, Hulsbergen-van der Kaa C, Oosterhof GO, VanderLaak JA, Kondacki H, Ruijs SH. Evaluation of chemotherapy in advanced urinary bladder cancer with fast dynamic contrast-enhanced MR imaging. Radiology. 1998 Jun;207(3):791-7. doi: 10.1148/radiology.207.3.9609906.
- [Background] Morgan B, Thomas AL, Drevs J, Hennig J, Buchert M, Jivan A, Horsfield MA, Mross K, Ball HA, Lee L, Mietlowski W, Fuxuis S, Unger C, O'Byrne K, Henry A, Cherryman GR, Laurent D, Dugan M, Marme D, Steward WP. Dynamic contrast-enhanced magnetic resonance imaging as a biomarker for the pharmacological response of PTK787/ZK 222584, an inhibitor of the vascular endothelial growth factor receptor tyrosine kinases, in patients with advanced colorectal cancer and liver metastases: results from two phase I studies. J Clin Oncol. 2003 Nov 1;21(21):3955-64. doi: 10.1200/JCO.2003.08.092. Epub 2003 Sep 29. PMID 14517187
- [Background] Tsuji M, Murota SI, Morita I. Docosapentaenoic acid (22:5, n-3) suppressed tube-forming activity in endothelial cells induced by vascular endothelial growth factor. Prostaglandins Leukot Essent Fatty Acids. 2003 May;68(5):337-42. doi: 10.1016/s0952-3278(03)00025-5. PMID 12711251
- [Derived] Al-Taan O, Stephenson JA, Spencer L, Pollard C, West AL, Calder PC, Metcalfe M, Dennison AR. Changes in plasma and erythrocyte omega-6 and omega-3 fatty acids in response to intravenous supply of omega-3 fatty acids in patients with hepatic colorectal metastases. Lipids Health Dis. 2013 May 7;12:64. doi: 10.1186/1476-511X-12-64. PMID 23648075